CLINICAL TRIAL: NCT01195337
Title: Social, Contextual, and Environmental Determinants of Physical Activity in Sedentary Minority Adults
Brief Title: Social Contextual Influences on Physical Activity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2008-0763
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Cancer; Prevention Harmful Effects
Keywords: Sedentary minority adult; Psychosocial factors; Environmental factors; Obesity; Physical Activity; PA; Cancer Risk; African Americans; Latino
MeSH Terms: conditions — Neoplasms; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Newsletters, Physical Activity (PA) Prescription Plan, Pedometer
  Interventions: Behavioral: PA Prescription Plan; Device: Pedometer; Behavioral: Newsletters

INTERVENTIONS:
Behavioral: PA Prescription Plan — Exercise program and instructions.
  Other Names: Physical Activity; Exercise
Device: Pedometer — Step monitor for individual PA progress.
Behavioral: Newsletters — 4 Newsletters with topics based on PA progression phases of adoption and maintenance.

SUMMARY:
The goal of this study is to learn why some black and Latino men and women choose not to exercise very often. Researchers also want to learn more about any social and environmental factors that may affect the way an exercise program is followed.

DETAILED DESCRIPTION:
If you chose to take part in this study, you will receive an exercise program, a pedometer, access to a social networking site, and newsletters to help you start becoming more physically active. A pedometer is a small device worn on the hip that counts the number of steps you have taken each day.

Study Visits:

You will come in for study visits 6 times while you are on study; 1 time at the beginning of the study called "screening", 1 time for an orientation visit 7 days after the screening visit, and for follow-up visits at 8, 26, 39, and 52 weeks after you begin the exercise program.

Baseline Tests:

If you are found to be eligible to take part on this study based on the results of the screening tests, the following tests and procedures will be performed:

* You will be asked to complete a computer-based survey. The questionnaires will ask questions about stress, your motivation for physical activity, any social support you may receive from others, the neighborhood you live in, and other physical activity-related topics. The questionnaires should take about 2 hours total to complete.
* Your blood pressure will be measured.
* Your height, weight, and waistline will be measured. To measure your waistline accurately, you may be asked to lift your shirt to expose your stomach area and to lower your pants to expose your mid-hip area. Waistline measurements will only take about 10 minutes to complete and will be performed in a private area.
* You will complete a fitness test. To complete the fitness test, you will either walk a circular path at the clinic for 6 minutes or complete a step test. The study staff will decide which test you will complete and will discuss the test with you in more detail. A study staff member will monitor you during this test.

Study Devices:

At the baseline visit, you will be given the following study devices:

* You will be given a smartphone to take home with you.
* You will fill out a set of questions on the smartphone each time you exercise. The questions will ask about the kind physical activity you are participating in, the location of where the physical activity is taking place, and the weather conditions outside. These questions will take about 1-2 minutes per day. Also, the smartphone will "beep" at random times (3 times per day) and set times (in the morning and evening) throughout the day to prompt you to answer a set of questions about your thoughts and feelings. The device will also automatically record your location using a Global Positioning System (GPS) during the time you are carrying the phone. This will take about 7-8 minutes per day. The research staff will call you 1 time each week to remind you to use the smartphone and will help with any smartphone problems that may occur. Each reminder phone call should last about 3 minutes. You will return the smartphone with you at the orientation visit for the study staff to download your answers.
* You will be given an accelerometer. You will wear the accelerometer for 7 days and then return it at the orientation study visit. An accelerometer is a small device that is worn on your hip that measures the amount of physical activity you do.

Orientation Study Visit:

At the orientation study visit, the following tests and procedures will be performed:

* You will be given a newsletter that contains information and strategies to help you start your exercise program.
* You will be given a smartphone again to take home.
* You will be given a physical activity (PA) prescription. The PA prescription outlines your exercise program and has instructions on the proper way to walk to decrease the chance of getting an injury. You will be instructed to start your PA prescription and carry the smartphone with you for 2 weeks. After 2weeks, you will return the smartphone by mail in a prepaid envelope that will be provided to you by the study staff.
* You will be given a pedometer to wear when you are ready to start your PA prescription.

Weeks 8, 26, 39, and 52 Study Visits:

For each of these study visits, the following tests and procedures will be performed:

* You will return the accelerometer at each visit for the study staff to review, and you will take it home at the end of each visit. The staff member will provide you with the device at your Week 8 visit and you will receive an envelope for return. The smartphone will also be given to you at Weeks 26 and 39, and you will be required to mail it back. For Week 52 you will receive the device 1 week before and return it at your Week 52 visit. You should tell a research staff member right away about any problems you may have using the smartphone.
* You will complete the computer-based survey.
* Your blood pressure will be measured.
* Your height, weight, and waistline will be measured.

You will receive phone calls between study visits to remind you to complete the questions on the smartphone.

At the Weeks 26 and 52 study visits, in addition to the tests and procedures listed above, you will complete the fitness test again and return the smartphone.

Length of Study:

You will remain in the study for up to 1 year. Your participation on this study will be over after you complete the study visit at Week 52.

Other Information:

You may be contacted by phone, mail, text messaging, and/or email at any time while you are taking part in this study to be reminded about the study visits. You will be asked to give the names and contact information of family members and/or friends for the study staff to contact in the event they cannot reach you first.

This is an investigational study.

Up to 300 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Black or Latino (self-defined by participant) ages 25-60 years
2. Currently sedentary, defined as self-reported physical activity of </=90 minutes per week over the past 6 months
3. Ready and physically able to start being physically active. Determined by asking participant if they intend to start being physically active within the next 30 days.
4. Have a home address where information can be mailed
5. Able to read English at a 6th grade level as assessed by the REALM
6. If uncontrolled hypertension or other physical limitations that might be aggravated by participation in lifestyle moderate-intensity physical activity as determined by PA Readiness Questionnaire (PAR-Q). Participants with BP readings >/=140/90mm Hg, will have to provide a doctors note or medical clearance.
7. Live within Harris County

Exclusion Criteria:

1. Pregnant or thinking about becoming pregnant during the study period
2. Another person in the same household is enrolled in the study
3. Physical limitation that prevents engaging in PA
4. MD Anderson employees who work in the Division of Cancer Prevention and Population Sciences

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 300 black or Latino participants in the greater Houston, Texas area.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2010-08-16 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Participant Physical Activity Outcome | 1 year
  Physical Activity (PA) outcome measured at four time points post baseline (weeks 8, 26, 39, and 52)

CONTACTS AND LOCATIONS:
Overall Officials: Lorna H. McNeill, PHD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org